CLINICAL TRIAL: NCT02601521
Title: Comparative Effectiveness of Two Tobacco Cessation Interventions for Employees of Partners HealthCare, Inc.
Acronym: PiHQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Partners HealthCare, Inc. (Industry)
Responsible Party: Principal Investigator, Nancy A. Rigotti, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000002/MGH
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Smoking Cessation; Tobacco Use Disorder
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internal coaching program (Experimental): The internal coaching program uses a chronic disease management strategy to treat tobacco use and dependence. The program provides evidence-based treatment consisting of up to 12 months of services from a tobacco coach based at Partners HealthCare. The tobacco coach offers (1) repeated smoking cessation counseling delivered by proactive telephone calls, emails, and interactive voice response [automated phone calls] and (2) facilitated access to a new Partners HealthCare Inc., health insurance benefit that provides access to all FDA-approved smoking cessation medications without copay or prior approval.
  Interventions: Behavioral: Internal tobacco coach
- External coaching program (Active Comparator): The external coaching program consists of referral to the Massachusetts Tobacco Control Program's Smokers Helpline, a free program offering multi-session proactive telephone counseling for 3 months to individuals who are ready to quit smoking. Individuals in this arm also receive information about Partners HealthCare, Inc.'s new health insurance benefit that provides access to all FDA-approved smoking cessation medications without copay or prior approval.
  Interventions: Behavioral: External tobacco coach

INTERVENTIONS:
Behavioral: Internal tobacco coach — The internal coaching program will provide cognitive-behavioral counseling and medication adherence support for smokers who are ready to quit in the next 3 months It consists of:
  1. Telephone counseling by the Tobacco Coach (8 calls over 12 weeks). supplemented by automated phone calls using interactive voice response. At each IVR contact, smokers can request a call back from the Tobacco Coach. Smokers who are not quit after 3 months can restart into the 12-week counseling program.
  2. The Tobacco Coach will assist smokers in choosing pharmacotherapy and in obtaining a prescription from the smoker's physician.
  3. Support and monitoring for 12 months using automated phone calls. If relapse occurs, the smoker will have the option to return to the active 12-week program.
  Arms: Internal coaching program
Behavioral: External tobacco coach — Referral to Massachusetts Smokers Helpline (telephone quitline operated by the Massachusetts Tobacco Control Program) for proactive telephone counseling.
  Arms: External coaching program

SUMMARY:
Specific Aim: To conduct a randomized controlled trial among permanent employees of Partners HealthCare, Inc., and their adult dependents, who are current tobacco smokers. The trial will compare two interventions designed to help smokers stop using tobacco: (1) External Coaching Program (Standard Care) and (2) Internal Coaching Program, a chronic disease management strategy for treating tobacco use and dependence.

ELIGIBILITY:
Inclusion Criteria:

* Current permanent employee of Partners Healthcare, Inc. or their adult dependent
* Current tobacco smoker (smoked a cigarette, even a puff, in the past 30 days)

Exclusion Criteria:

* Temporary, per diem or former employee of Partners Healthcare, Inc.
* Plan to leave Partners employment in the next 12 months
* Inability to give informed consent or participate in counseling due to serious psychiatric disorder or cognitive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Tobacco abstinence for the past 30 days | 6 months after enrollment

SECONDARY OUTCOMES:
Tobacco abstinence for the past 30 days | 3 months after enrollment
Tobacco abstinence for the past 30 days | 12 months after enrollment
Quit attempt | Intentional tobacco abstinence for at least 24 hours since enrollment

OTHER OUTCOMES:
Duration of use of tobacco cessation pharmacotherapy | at 3 months and at 6 months after enrollment
  Includes any FDA-approved product (nicotine patch, gum, lozenge, inhaler, nasal spray or bupropion or varenicline
Smoking cessation counseling contacts | at 3 months and at 6 months after enrollment
  Number of telephone calls with an internal or external tobacco coach to address smoking cessation

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States